CLINICAL TRIAL: NCT06775704
Title: Résultats Cliniques et Radiologiques du Dispositif de resurfaçage de Hanche ROMAXTM Medacta
Brief Title: Clinical and Radiological Outcomes of the ROMAX Hip Resurfacing System
Status: Recruiting | Type: Observational
Sponsor: Medacta International SA (Industry)
Responsible Party: Sponsor
Other Study IDs: P 01.012.07
Record Dates: First submitted 2025-01-09; First posted 2025-01-15 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Arthritis (Hip); Hip Dysplasia, Congenital
Keywords: resurfacing
MeSH Terms: conditions — Arthritis; Hip Dislocation, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ROMAX: Patients undergoing hip resurfacing surgery with ROMAX system
  Interventions: Device: Hip resurfacing system

INTERVENTIONS:
Device: Hip resurfacing system — Hip resurfacing with ROMAX system

SUMMARY:
The goal of this observational study is to collect clinical and radiological data to monitor the safety and performance of the ROMAX hip resurfacing system. The main parameter that will be measured is the rate of revisions at 10 years.

DETAILED DESCRIPTION:
This single-center, post-market, prospective, longitudinal, and uncontrolled cohort study aims to evaluate the survival rate of the Medacta ROMAX hip resurfacing system, particularly focusing on dislocations and the potential consequences of wear over a 10-year period. Additionally, the study will assess clinical performance through patient-reported outcomes (PROMs) and analyze the migration behavior of the device using the CTMA method in a subgroup of 40 patients. The study will include a total of 150 cases, with 40 patients undergoing CTMA analysis at 3 years post-surgery. Eligible patients will be informed during preoperative visits and included upon signing the consent form, prior to surgery. Participation in the CTMA subgroup is optional and does not affect overall study inclusion. Follow-ups will be conducted at 3 months, 1, 3, 5, and 10 years. Data collection will include clinical scores, clinical and radiological data related to preoperative and postoperative status, and perioperative surgical details.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for hip resurfacing, suitable for the implantation of a Medacta ROMAX hip resurfacing system according to the manufacturer's defined indication for use.
* Aged between 18 and 65 years at the time of surgery.
* Ability and willingness to provide written informed consent for participation.

Exclusion Criteria:

* Active infection
* BMI > 40
* Mental illness, when the known pathology is likely to compromise the patient's ability to consent, affect the patient's assessment of their progress, or complete follow-up appointments and exams.
* Significantly deformed anatomy (at the surgeon's discretion)
* Osteomalacia where the fixation of an uncemented implant is contraindicated
* Active rheumatoid arthritis
* Osteoporosis
* Metabolic disorders likely to impair bone formation and for which the fixation of an uncemented implant is contraindicated
* Muscle atrophy or neuromuscular disease
* Known allergy or hypersensitivity to the implant material
* Any patient who cannot or does not wish to give informed consent to participate in the study
* Patients whose chances of regaining independent mobility would be compromised by known concomitant medical issues.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 150 patients undergoing hip resurfacing surgery and receiving the ROMAX system will be recruited consecutively by the study investigator. All patients will be offered to join the CTMA subgroup until the number of 40 subjects is reached. Choosing not to participate in the CTMA subgroup will not prevent the patient from participating in the study.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2037-04-01 (Estimated); Study Completion 2037-04-01 (Estimated)

PRIMARY OUTCOMES:
Implant survival | 10 years
  Survival of the implant through Kaplan-Meier analysis based on revisions

SECONDARY OUTCOMES:
Harris Hip Score (HHS) | 3 months, 1 year, 3 years, 5 years, 10 years
  Measure of dysfunction ranging from 0 to 100, where higher values represent better outcomes.
Forgotten Joint Score (FJS) | 3 months, 1 year, 3 years, 5 years, 10 years
  Patient-reported outcome measure that evaluates joint dysfunction. It ranges from 0 to 100, with higher scores indicating better outcomes
Postel-Merle d'Aubigné Score (PMA) | 3 months, 1 year, 3 years, 5 years, 10 years
  Clinical rating system used to assess hip function. It ranges from 0 to 18, with higher scores indicating better hip function and fewer limitations in activities.
Oxford Hip Score (OHS) | 3 months, 1 year, 3 years, 5 years, 10 years
  Patient-reported outcome measure designed to assess hip function and pain. It ranges from 0 to 48, with higher scores indicating better function and less pain.
UCLA Activity Scale | 3 months, 1 year, 3 years, 5 years, 10 years
  Questionnaire assessing physical activity level from 1 (low) to 10 (high).
HOOS (Hip injury and Osteoarthritis Outcome Score) Symptoms subscale | 3 months, 1 year, 3 years, 5 years, 10 years
  Patient-reported outcome measure comprising 5 questions assessing hip joint symptoms and stiffness. It ranges from 0 to 100, with higher values indicating better outcomes.
Radiologic Evaluation | 3 months, 1 year, 3 years, 5 years, 10 years
  Assessment of implant positioning and radiographic appearence.
CT-micromotion analysis (CTMA) | 3 months, 1 year, 3 years
  CT-based evaluation of implant movement and wear. Will be performed on a subgroup of patients (40)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de Lille, Lille, France

IPD SHARING:
Plan to Share IPD: No